CLINICAL TRIAL: NCT03461614
Title: Effects of Core Stabilization Exercises on Pulmonary Functions, Respiratory Muscle Strength and Functional Capacity in Adolescents With Substance Use Disorder. A Randomized Controlled Study
Brief Title: Effects of Core Stabilization Exercises on Pulmonary Functions, Respiratory Muscle Strength and Functional Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, RUSTEM MUSTAFAOGLU, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Substance Use Disorders; Substance Abuse; Substance Use
Keywords: pulmonary function; respiratory muscle strength; functional capacity; core exercises; rehabilitation
MeSH Terms: conditions — Substance-Related Disorders | interventions — Control Groups; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): In addition to the service routine rehabilitation program, in this group all participant receive as group training with instructor supervising 5-6 participants. The specific days of the week and time of day in which the participants trained remained constant throughout each training protocol. Training programs lasted 6 weeks and comprised 2 training sessions per week with a total of 12 training sessions. A 45-60 min training sessions per week with a 2 day gap between each session.
  Interventions: Other: Exercise group
- Control Group (Other): In addition to the service routine rehabilitation program, participants in the Control group participated in leisure activities such as table tennis/basketball under service staff supervision for 45-60 minutes, 2 times a week, 6 weeks similar time period of Exercise group.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Exercise group — Exercise group mainly conducted the 5 core stabilization exercises as described by McGill. These include the curl-up, side bridge, trunk extension, double leg lifts and bird-dog exercises that support respiratory functions. In other words, every single training session consisted of frontal, dorsal, and lateral core exercise. In general, participants always exercised in group so that for integration and motivation. During training weeks 1-2, participants exercises with 3 sets per exercise and 10 s contraction time and 10 repetitions. During training weeks 3-4, contraction times and repetitions were increased to 15 s and 15 repetitions. Additionally, increasing the complexity of exercises, adding opposite limb movements and increasing the lever arm of the exercises were done.
  Other Names: Core stabilization exercise
  Arms: Exercise Group
Other: Control group — In addition to the service routine rehabilitation program mentioned above, participants in the Control group participated in leisure activities such as table tennis/basketball under service staff supervision for 45-60 minutes, 2 times a week, 6 weeks similar time period of Exercise group.
  Other Names: Aerobic exercise
  Arms: Control Group

SUMMARY:
In recent years adolescent substance abuse is a serious and growing problem. Substance use among adolescents means the use of alcohol, opiates, amphetamines, inhalants, cocaine, marijuana, benzodiazepines, hallucinogens, and anabolic steroids. The United Nations Office on Drugs and Crime reports that approximately 5% of the world's population used an illicit drug in 2010 and it is estimated that heroin, cocaine and other drugs are responsible for 0.1 to 0.2 million deaths per year.

There is a limited number of studies in the literature that investigate the relationship between substance use disorder and respiratory functions. In Taylor et al., study reported that the proportion of cannabis-dependent study members with an FEV1/FVC ratio of, 80% was 36% compared to 20% for non-smokers. Another research of Taylor et al., in longitudinal observations over 8 years in young adults (cannabis smoking on lung function in young adults between the ages of 18 and 26) revealed a dose-dependent relationship between cumulative cannabis consumption and decline in FEV1/VC. In a monograph, stated that follow-up studies of regular cannabis-only smokers also found impaired respiratory function and pathological changes in lung tissue like those preceding the development of chronic obstructive pulmonary disease .

The core anatomically described as a box, with the abdominals at the front, spinal and gluteal muscles at the back, the diaphragm on the top, and the pelvic floor and hip muscles on the bottom. Correct breathing is vital to abdominal training because respiratory muscles are directly involved during common core stability exercises. Moreover, the diaphragm, a component of core stability, plays a role in respiration and trunk stability by controlling intra-abdominal pressure . Oh et al.reported that, 30-min, 3 days a week for 8 weeks lumbar stabilization exercise had a more positive effect on pulmonary function than general physical therapy on stroke patients.

Our hypothesis was that core exercises may positive effect on respiratory functions and functional capacity of substance use disorder individuals. The aim of our study is to investigate the effects of core exercises on respiratory functions and functional capacity in adolescents with substance use disorder.

DETAILED DESCRIPTION:
Subjects: The study sample comprised of 15-18 year old male. Participants were required to be in-residence at the treatment center and meet Diagnostic and Statistical Manual-V criteria for substance use disorder in Mental Health and Neurological Diseases Training and Research Hospital for Psychiatry, Neurology and Neurosurgery; Child and Adolescent Drug and Alcohol Dependence Treatment Center (CEMATEM) in Istanbul.

Sample Size Determination: The sample size and power calculations were performed using the Instat sample size calculator. The calculations were based on the average value of the 6-Minute Walk Test in the 15-20 age group was 725.8 meters and the standard deviation (SD) was 61.2 meters (28), in the 95% confidence interval, an alpha level of 0.05, a β level of 5% and a power of 95%.These parameters generated a sample size of at least 18 participants for each group.

Randomization Study Protocol: The participants were randomly assigned to 1 of 2 parallel groups to receive either Exercise or Control. To allocate the participants to the groups, using the method of randomly permuted blocks using Research Randomizer, a program published on a publicly accessible official website (www.randomizer.org). Computerized random numbers were conducted, and sequentially numbered index cards with the random assignment were prepared. The index cards were folded and placed in sealed, opaque envelopes. Then, the investigator opened each envelope and allocated the participants to the Exercise or control group according to the selected index card.

ELIGIBILITY:
Inclusion Criteria:

* were between 15 and 18 years of age,
* met current Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for substance use disorder,
* be using substances over a year,
* have not participated regularly in any exercise training program for the past six months,
* were currently engaged in inpatient substance abuse treatment.

Exclusion Criteria:

* a history of psychotic disorder or current psychotic symptoms,
* physical disabilities or medical problems,
* inability to adapt to the evaluation and treatment program,
* have a respiratory system problems such as bronchiectasis, asthma and tuberculosis, infectious health problem (HIV, hepatitis B etc.).

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test | 6 weeks
  Pulmonary functions were measured using portable spirometry (Spirobank II; Medical International Research Rome, Italy). Measurements were performed according to the criteria of the American Thoracic Society (ATS) and the European Respiratory Society (ERS) guidelines.
Maximal Inspiratory and Expiratory Pressures | 6 weeks
  Participants' maximal inspiratory and expiratory pressures was measured and recorded according to ATS/ERS criteria using a portable, electronic intraoral pressure gauge (Carefusion, USA) . During the test, subjects were encouraged verbally. Technically acceptable, the highest of at least three measurements that did not differ by more than 5 cm H2O was recorded for maximal inspiratory and expiratory pressures. A percentages of the predicted values of maximal inspiratory and expiratory pressures were expressed as described by Black and Hyatt.
Functional Capacity | 6 weeks
  Functional capacity was measured with the 6-Minute Walk Test (6MWT) according to the guideline of ERS. The 6MWT to be a reliable, reproducible, and valid functional test for assessing exercise tolerance and endurance. Subjects were instructed to walk from one end to the other of a 30 m hallway at their own pace, while attempting to cover as much ground as possible in the allotted 6 min. The test was self-paced and the subject could rest if he or she so wished.

SECONDARY OUTCOMES:
Respiratory Related Symptoms | 6 weeks
  Respiratory related symptoms were assessed by using the respiratory section of the third National Health Nutrition Examination Survey (NHANES III) and the Medical Research Council breathlessness questionnaire were used to record reported respiratory symptoms. Questionnaires were given as face-to-face interviews by one investigator in a standardised manner.
The Modified Medical Research Council (mMRC) Dyspnoea Scale | 6 weeks
  The Medical Research Council (MRC) dyspnoea scale has been in use for many years for grading the effect of breathlessness on daily activities. This scale actually measures perceived respiratory disability, the World Health Organization definition of disability being "any restriction or lack of ability to perform an activity in the manner or within the range considered normal for a human being". The MRC dyspnoea scale is simple to administer as it allows the patients to indicate the extent to which their breathlessness affects their mobility. The person indicates the degree of breathlessness with a score of 0-4. Level 0 refers to there is not breathless, level 4 refers to there is a severe breathless.
The Fagerstrom Test of Nicotine Dependence (FTND) | 6 weeks
  The FTND is a widely used 6-item scale with high test-retest validity. The nicotine dependence of the total score obtained from the test,low (0-3 points), moderate (4-6 points) and high (≥7 points).

CONTACTS AND LOCATIONS:
Overall Officials: Rustem Mustafaoğlu, PT, Principal Investigator — İstanbul Üniversitesi, Sağlık Bilimleri Fakültesi
Locations (1):
- Rustem Mustafaoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Carney T, Myers BJ, Louw J, Okwundu CI. Brief school-based interventions and behavioural outcomes for substance-using adolescents. Cochrane Database Syst Rev. 2014 Feb 4;(2):CD008969. doi: 10.1002/14651858.CD008969.pub2. PMID 24563456
- [Result] Chakravarthy B, Shah S, Lotfipour S. Adolescent drug abuse - awareness & prevention. Indian J Med Res. 2013 Jun;137(6):1021-3. No abstract available. PMID 23852281
- [Result] Taylor DR, Poulton R, Moffitt TE, Ramankutty P, Sears MR. The respiratory effects of cannabis dependence in young adults. Addiction. 2000 Nov;95(11):1669-77. doi: 10.1046/j.1360-0443.2000.951116697.x. PMID 11219370
- [Result] Taylor DR, Fergusson DM, Milne BJ, Horwood LJ, Moffitt TE, Sears MR, Poulton R. A longitudinal study of the effects of tobacco and cannabis exposure on lung function in young adults. Addiction. 2002 Aug;97(8):1055-61. doi: 10.1046/j.1360-0443.2002.00169.x. PMID 12144608
- [Result] Key J. 'The core': understanding it, and retraining its dysfunction. J Bodyw Mov Ther. 2013 Oct;17(4):541-59. doi: 10.1016/j.jbmt.2013.03.012. Epub 2013 Jun 28. PMID 24139017
- [Result] Park SJ, Lee JH, Min KO. Comparison of the effects of core stabilization and chest mobilization exercises on lung function and chest wall expansion in stroke patients. J Phys Ther Sci. 2017 Jul;29(7):1144-1147. doi: 10.1589/jpts.29.1144. Epub 2017 Jul 15. PMID 28744034
- [Result] Oh DS, Park SE. The effect of lumbar stabilization exercise on the pulmonary function of stroke patients. J Phys Ther Sci. 2016 Jun;28(6):1896-900. doi: 10.1589/jpts.28.1896. Epub 2016 Jun 28. PMID 27390442
- [Result] Macleod J, Robertson R, Copeland L, McKenzie J, Elton R, Reid P. Cannabis, tobacco smoking, and lung function: a cross-sectional observational study in a general practice population. Br J Gen Pract. 2015 Feb;65(631):e89-95. doi: 10.3399/bjgp15X683521. PMID 25624312
- [Result] Fletcher C. Standardised questionnaire on respiratory symptoms: a statement prepared and approved by the MRC Committee on the Aetiology of Chronic Bronchitis (MRC breathlessness score). Bmj. 1960;2(2):1665.
- [Result] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Result] Stavem K, Rogeberg OJ, Olsen JA, Boe J. Properties of the Cigarette Dependence Scale and the Fagerstrom Test of Nicotine Dependence in a representative sample of smokers in Norway. Addiction. 2008 Sep;103(9):1441-9. doi: 10.1111/j.1360-0443.2008.02278.x. PMID 18783499
- [Result] Fagerstrom KO. Measuring degree of physical dependence to tobacco smoking with reference to individualization of treatment. Addict Behav. 1978;3(3-4):235-41. doi: 10.1016/0306-4603(78)90024-2. No abstract available. PMID 735910
- [Result] Uysal MA, Kadakal F, Karsidag C, Bayram NG, Uysal O, Yilmaz V. Fagerstrom test for nicotine dependence: reliability in a Turkish sample and factor analysis. Tuberk Toraks. 2004;52(2):115-21. PMID 15241694
- [Result] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Result] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Result] Domenech-Clar R, Lopez-Andreu JA, Compte-Torrero L, De Diego-Damia A, Macian-Gisbert V, Perpina-Tordera M, Roques-Serradilla JM. Maximal static respiratory pressures in children and adolescents. Pediatr Pulmonol. 2003 Feb;35(2):126-32. doi: 10.1002/ppul.10217. PMID 12526074
- [Result] Puente-Maestu L, Palange P, Casaburi R, Laveneziana P, Maltais F, Neder JA, O'Donnell DE, Onorati P, Porszasz J, Rabinovich R, Rossiter HB, Singh S, Troosters T, Ward S. Use of exercise testing in the evaluation of interventional efficacy: an official ERS statement. Eur Respir J. 2016 Feb;47(2):429-60. doi: 10.1183/13993003.00745-2015. Epub 2016 Jan 21. PMID 26797036
- [Result] Flemmen G, Unhjem R, Wang E. High-intensity interval training in patients with substance use disorder. Biomed Res Int. 2014;2014:616935. doi: 10.1155/2014/616935. Epub 2014 Mar 2. PMID 24724089
- [Result] Buchowski MS, Meade NN, Charboneau E, Park S, Dietrich MS, Cowan RL, Martin PR. Aerobic exercise training reduces cannabis craving and use in non-treatment seeking cannabis-dependent adults. PLoS One. 2011 Mar 8;6(3):e17465. doi: 10.1371/journal.pone.0017465. PMID 21408154